CLINICAL TRIAL: NCT06303102
Title: Effects of Segmental and Pursed Lip Breathing Exercises on Neck Pain, Functional Disability and Quality of Life in Upper Cross Syndrome
Brief Title: Effects of Segmental and Pursed Lip Breathing Exercises on Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0356
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: UPPER CROSS SYNDROME
Keywords: Breathing Exercises; Cervical Pain; Disability; Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental Group A (Manual PT/ Conventional PT Treatment + Segmental and Pursed Lip Breathing Exercise)
  Interventions: Other: Manual PT/ Conventional PT Treatment + Segmental and Pursed Lip Breathing Exercise
- Controlled (Other): Group B (Manual PT/Conventional PT Treatment)
  Interventions: Other: Manual PT/Conventional PT Treatment

INTERVENTIONS:
Other: Manual PT/ Conventional PT Treatment + Segmental and Pursed Lip Breathing Exercise — 20 patients will receive conventional physical therapy treatment (hot pack, electrical stimulation, myofascial release, ROM and strengthening exercises) along with segmental and pursed lip breathing exercises.
  Arms: Experimental
Other: Manual PT/Conventional PT Treatment — 20 patients will receive conventional physical therapy treatment (hot pack, electrical stimulation, myofascial release, ROM and strengthening exercises).
  Arms: Controlled

SUMMARY:
Upper cross syndrome is relative prevalent 67% musculoskeletal disorder among general population due to increased usage of smart gadgets and poor postural habits. Upper cross syndrome is known for initiating malfunction of cervical and upper back muscles also associated with respiration. Individuals with upper cross syndrome may present with relaxed supine positioning, they may having normal respiratory mechanics but might be converted to accessory muscles activated pattern. Neck pain is the most common type of pain in non-traumatic conditions, affecting about 75.7% of people. The aim of this study is to compare the effects of segmental and pursed lip breathing exercises on pain, functional disability and quality of life in population with upper cross syndrome.

Current study will be randomized controlled trial conducted at Ismail Medicare Jhang, 40 patients according to inclusion criteria will be included in the study. They will be allocated into 2 groups by non-probability purposive sampling technique. Group A (control group) will receive conventional physical therapy treatment (hot pack, electrical stimulation, myofascial release, ROM and strengthening exercises) while Group B (experimental group) receive conventional physical therapy treatment with segmental and pursed lip breathing exercises. Outcome measures are Pain Numeric Scale, Quality of life (SF 36) and Functional disability (neck disability index). These tools will measure neck function and neck pain intensity. Treatment time will be 4 weeks, 3 sessions per week, each session will be 45 minutes long, and measurements will be taken after 4 weeks. Data will be analyzed by SPSS version 25. After assessing normality of data by Shapiro - wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups analysis.

Key Words: Breathing Exercises, Cervical Pain, Disability, Upper Cross

ELIGIBILITY:
Inclusion Criteria:

* Both Gender >25-40 years
* Diagnosed with Upper Cross Syndrome, having neck pain intensity more than 5 on numeric pain rating scale and having pain from more than 3 months
* Positive Janda cervical flexion Test

Exclusion Criteria:

* Patient with other musculoskeletal disorder e.g cervicogenic headache excluded
* Neck pain with whiplash or headache disorder were not included
* Patients had any history of previous head and neck surgery excluded
* Any history of Infection in the cervical spine were not included
* Trigger points of trapezius were excluded

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
NPRS | 4 Weeks
  An outcome measure used to gauge adult pain intensity is the Numeric Pain Rating Scale (NPRS). "No pain" is represented by a score of '0' on the11-point numeric scale, while "pain as bad as you can imagine" or "worst pain imaginable" are represented by a score of '10'. An 11-point numerical scale goes from '0', which indicates no discomfort, to 10 symbolizing the most excruciating agony conceivable. Pre-post readings will be taken
Quality of Life (SF-36 questionnaire) | 4 Weeks
  The Short Form Survey (SF-36) is a tool used to measure various aspects of quality of life, such as body pain, physical well-being or functionality. Restrictions on role performance brought on by issues with one's physical, mental, or social well-being as well as one's general sense of health. Pre-post readings will be taken.
Neck Disability Index (NDI) | 4 Weeks
  The Oswestry Low Back Pain Disability Index was modified to create the Neck Disability Index (NDI). The purpose of this questionnaire is to gather information on how your neck pain has impacted your day-to-day functioning. The NDI is now a commonly used tool to assess neck pain-related self-rated disability. All ten items have a score ranging from 0 to 5. The purpose of this questionnaire is to gather information on how your neck pain has impacted your day-to-day functioning. The NDI is now a commonly used tool to assess neck pain-related self-rated disability. All ten items have a score ranging from 0 to 5. Pre-post readings will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Muriam Ghani, MSCPPT, Principal Investigator — Ripha International University-LHR
Locations (1):
- Ismail Medicare, Jhang, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baradaran Mahdavi S, Riahi R, Vahdatpour B, Kelishadi R. Association between sedentary behavior and low back pain; A systematic review and meta-analysis. Health Promot Perspect. 2021 Dec 19;11(4):393-410. doi: 10.34172/hpp.2021.50. eCollection 2021. PMID 35079583
- [Background] Csepregi E, Gyurcsik Z, Veres-Balajti I, Nagy AC, Szekanecz Z, Szanto S. Effects of Classical Breathing Exercises on Posture, Spinal and Chest Mobility among Female University Students Compared to Currently Popular Training Programs. Int J Environ Res Public Health. 2022 Mar 21;19(6):3728. doi: 10.3390/ijerph19063728. PMID 35329415
- [Background] de-la-Iglesia L, Bravo C, Rubi-Carnacea F. Upper crossed syndrome in secondary school students: A mixed-method study. J Taibah Univ Med Sci. 2023 Jan 24;18(4):894-907. doi: 10.1016/j.jtumed.2023.01.008. eCollection 2023 Aug. PMID 36852233
- [Background] Ghan GM, Babu VS. Immediate Effect of Cervico-thoracic Mobilization on Deep Neck Flexors Strength in Individuals with Forward Head Posture: A Randomized Controlled Trial. J Man Manip Ther. 2021 Jun;29(3):147-157. doi: 10.1080/10669817.2020.1834321. Epub 2020 Oct 22. PMID 33090945
- [Background] Arshadi R, Ghasemi GA, Samadi H. Effects of an 8-week selective corrective exercises program on electromyography activity of scapular and neck muscles in persons with upper crossed syndrome: Randomized controlled trial. Phys Ther Sport. 2019 May;37:113-119. doi: 10.1016/j.ptsp.2019.03.008. Epub 2019 Mar 21. PMID 30928841
- [Background] Mujawar JC, Sagar JH. Prevalence of Upper Cross Syndrome in Laundry Workers. Indian J Occup Environ Med. 2019 Jan-Apr;23(1):54-56. doi: 10.4103/ijoem.IJOEM_169_18. PMID 31040591